CLINICAL TRIAL: NCT00004344
Title: Purification of Testis-Stimulating Factor in Precocious Puberty
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11903; OHSU-3328
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: Precocious Puberty
Keywords: endocrine disorders; precocious puberty; rare disease
MeSH Terms: conditions — Puberty, Precocious; Endocrine System Diseases; Rare Diseases | interventions — Leuprolide; Testosterone

INTERVENTIONS:
Drug: leuprolide
Drug: testosterone

SUMMARY:
OBJECTIVES:

Purify and characterize a testis-stimulating factor in the blood of adult volunteers who had precocious puberty as boys.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Subjects are treated for 2 months with depot injections of leuprolide acetate every 4 weeks and testosterone replacement every 2 weeks. Hormone levels are tested every other week.

If luteinizing hormone and follicular-stimulating hormone levels are at or below detection on day 56, blood is drawn for a testis-stimulating factor bioassay and subsequent factor purification and characterization.

Volunteers are asked to repeat this 2-month procedure no more than 2 times every 12 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Adult men diagnosed with precocious puberty (familial testotoxicosis) as boys

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Barry Albertson, Study Chair — Oregon Health and Science University